CLINICAL TRIAL: NCT00153361
Title: Project Mix: Behavioral Intervention to Reduce Sexual Risk Behavior of Substance-Using (Non-Injection) Men Who Have Sex With Men
Brief Title: Project MIX: Behavioral Intervention to Reduce Risk Among Substance-Using MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gordon Mansergh (U.S. Federal Agency)
Collaborators: New York Blood Center (Other); San Francisco Department of Public Health (Other Government); University of Illinois at Chicago (Other); Health Research Association (Other)
Responsible Party: Sponsor-Investigator, Gordon Mansergh, Project Officer/Senior Scientist, Centers for Disease Control and Prevention
Organization: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-3985; U65/CCU522209; U65/CCU922215; U65/CCU222309; U65/CCU922213
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Intervention (Experimental): Behavioral discussion sessions focused on reducing substance use and sexual risk behavior
  Interventions: Behavioral: Discussion Group
- Comparison (Active Comparator): Video discussion on health issues unrelated to HIV prevention and substance use
  Interventions: Behavioral: Video Discussion Group
- Control (No Intervention): Waitlist control

INTERVENTIONS:
Behavioral: Discussion Group
  Arms: Intervention
Behavioral: Video Discussion Group
  Arms: Comparison

SUMMARY:
The purpose of this project is to test the efficacy of an HIV prevention behavioral intervention to reduce sexual risk for HIV infection among non-injection, substance-using men who have sex with men (SUMSM). The primary goal of the intervention is to reduce HIV transmission by reducing the incidence of unprotected anal sex while under the influence of alcohol and other drugs (AOD).

DETAILED DESCRIPTION:
Men who have sex with men (MSM) continue to be the largest risk category for incident and prevalent cases of HIV and AIDS in the U.S. Studies of MSM have established an association between alcohol and other drug (AOD) use and risky sexual behaviors. Although studies have assessed and confirmed the association of AOD use and unsafe sex, few have focused specifically on reducing sexual risk of SUMSM.

Sexual risk reduction interventions for MSM identified in the published scientific literature have demonstrated that they are generally effective at reducing sexual risk behaviors among MSM. However, none of these interventions specifically targeted non-injecting SUMSM. Thus, a gap exists in prevention efforts to reduce HIV transmission among SUMSM.

The primary aim of the Project Mix overall is to develop and evaluate a practical intervention strategy that is specifically tailored to the needs of non-injecting SUMSM. The intent of the intervention is to decrease the number of unprotected anal sex partners (and acts) while under the influence of AOD and in general.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years of age or older;
* self-identify as male;
* understand and read English;
* live within the metropolitan area;
* report being drunk or "buzzed" on alcohol 2 or more times or high on non-injection drugs at least once during (or two hours before) anal sex in the past six months;
* have had at least one unprotected anal sex episode in the past six months with a male partner of unknown or different HIV-status than their own (i.e., DUA)

Exclusion Criteria:

* report only marijuana, only Viagra or only marijuana and Viagra use during anal sex (current research shows that marijuana use is not associated with sexual risk behavior);
* report injecting drugs (eligible if only methamphetamine, steroids, hormones and/or prescribed medications) in the past six months;
* have known their HIV-positive status for less than six months (this is done to allow for psychological and behavioral adjustment following an initial HIV diagnosis and this time frame coincides with our screening window); these men (if they so desire) will be put on a wait list and contacted after 6 months have passed since their first HIV-positive test result;
* are currently involved in another HIV behavioral intervention study for MSM [local study site identifies a list of such studies in their community at the time of the trial];
* have a specific plan to move from the metropolitan area within the next 15 months;
* participated in the pilot phase of the project;
* other reasons that the investigators deem would make participation either detrimental to the participant or to the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1686 (Actual)
Dates: Start 2002-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Decrease in the number of unprotected anal sex partners (and acts) while under the influence of AOD as reported at 3-, 6-, and 12-month follow-up assessments compared to baseline assessments. | 3 months
Decrease in the number of unprotected anal sex partners (and acts) as reported at 3-, 6-, and 12-month follow-up assessments compared to baseline assessments. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Mansergh, PhD, Principal Investigator — Centers for Disease Control and Prevention
Locations (6):
- United States (6):
  - Health Research Association, Hollywood, California
  - San Francisco Department of Public Health, San Francisco, California
  - The University of Illinois at Chicago, Chicago, Illinois
  - Howard Brown Health Center, Chicago, Illinois
  - New York Blood Center, New York, New York
  - Project Achieve, New York, New York

REFERENCES:
- [Derived] Mansergh G, Koblin BA, McKirnan DJ, Hudson SM, Flores SA, Wiegand RE, Purcell DW, Colfax GN; Project MIX Study Team. An intervention to reduce HIV risk behavior of substance-using men who have sex with men: a two-group randomized trial with a nonrandomized third group. PLoS Med. 2010 Aug 24;7(8):e1000329. doi: 10.1371/journal.pmed.1000329. PMID 20811491